CLINICAL TRIAL: NCT06889870
Title: PECS II Blockade vs. Local Anesthesia: Postoperative Pain Control in Opioid-Free Oncologic Breast Surgery
Brief Title: Evaluating The Efficacy Of Pecs II Blockade Compared To Local Anesthetic Infiltration In Controlling Postoperative Pain In Patients Undergoing Oncologic Breast Surgery Under Opioid Free/Sparing Anesthesia.
Acronym: pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas de Minas Gerais (Other)
Responsible Party: Principal Investigator, Alessandra Hubner de Souza, Main supervisor of the study, statistical analyst and specialist in pain studies; pHd IN pHARMACOLOGICAL SCIENCES, Faculdade de Ciências Médicas de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FCMMG
Record Dates: First submitted 2024-12-19; First posted 2025-03-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Pain; Pain Management; Anesthesia
Keywords: ANESTHESIA; BREAST NEOPLASMS; NERVE BLOCK; OPIOID ANALGESICS
MeSH Terms: conditions — Pain; Agnosia; Breast Neoplasms | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
  - both the researcher and those taking part in the study do not know which intervention each participant is receiving is receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anesthetic infiltration at the surgical incision site group (LOC group) (Active Comparator): In the LOC group, local infiltration will be carried out by the surgeon before the surgical incision. Adrenaline 1:20000 will be added to the anesthetic solution in the LOC group for the surgeon's convenience in order to better control perioperative bleeding
  Interventions: Procedure: Local Anesthesia
- PECS II blockade (PEC group) (Experimental): In the PEC group, the PECS II block will be performed by the same anesthesiologist and will be performed before the skin incision, using the technique described by Blanco at al, 2012. A 10 ml solution of ropivacaine (0.3%) will be administered into the fascia between the pectoralis major and pectoralis minor muscles and 20 ml of the same anesthetic solution between the pectoralis minor and serratus muscles.
  Interventions: Procedure: Pectoral Nerve Block

INTERVENTIONS:
Procedure: Pectoral Nerve Block — In the PEC group, the PECS II block will be performed by the same anesthesiologist and will be performed before the skin incision, using the technique described by Blanco at al, 2012. 10 ml of ropivacaine solution (0.3%) will be administered into the fascia between the pectoralis major and pectoralis minor muscles and 20 ml of the same anesthetic solution between the pectoralis minor and serratus muscles.
  Arms: PECS II blockade (PEC group)
Procedure: Local Anesthesia — In the LOC group, local infiltration will be carried out by the surgeon before the surgical incision. Adrenaline 1:20000 will be added to the anesthetic solution in the LOC group for the surgeon's convenience in order to better control per operative bleeding. In the PEC group, a solution of adrenaline in the same concentration in 0.9% saline will be infiltrated, also just to control bleeding in the surgical field.
  Arms: anesthetic infiltration at the surgical incision site group (LOC group)

SUMMARY:
Breast cancer is the malignant neoplasm with the highest incidence in women in Brazil, with the exception of non-melanoma skin tumors. Breast cancer surgery is an important part of treatment and post-operative pain needs to be adequately prevented and treated. This prospective, randomized, double-blind clinical study aims to evaluate the efficacy of interfascial pectoral nerve block (PECS II) compared to local anesthetic infiltration at the surgical site in patients undergoing breast cancer surgery in terms of pain and nausea. Data collection will be carried out at the Nossa Senhora das Dores Hospital with 133 patients, who will be divided into two groups: the PEC group will undergo PECS II blockade and the LOC group will undergo local anesthetic infiltration at the surgical site. Both interventions will be performed after the induction of opioid-free/sparing balanced general anesthesia. At the end of surgery, the patients will be taken to the post-anesthetic recovery room (PACU), where post-operative pain will be monitored on arrival and at 30-minute intervals up to two hours after surgery, and before the patient is discharged the following day. A visual analog scale (VAS) will be used, and PONVs will also be recorded. After a 2-hour stay in the PACU, they will be transferred to the ward, and after 24 hours, they will be reassessed using the same parameters. Opioid consumption will be recorded in the PACU and during hospitalization, as well as the occurrence of nausea or vomiting and compared between the groups, and side effects and complications will be monitored.

DETAILED DESCRIPTION:
Introduction:

Breast cancer is the most prevalent malignant neoplasm among women in Brazil, and oncologic surgery is an essential part of its treatment. Postoperative pain is a significant challenge, especially in approaches with general anesthesia. Methods such as PECS II blockade and infiltration of local anesthetics have been used for pain management and reduction of opioid consumption.

Objective:

The study aims to evaluate the effectiveness of the PECS II interfascial block in comparison with local anesthetic infiltration in controlling postoperative pain in patients undergoing breast oncology surgery under general anesthesia with minimal use of opioids (opioid-free/sparing).

Methodology:

This is a prospective, randomized, double-blind clinical trial involving 133 patients. They will be divided into two groups:

PEC group: will receive the PECS II block; LOC group: will be treated with local anesthetic infiltration at the surgical site.

Both interventions will take place after induction of anesthesia. The outcomes assessed include postoperative pain (using a visual analog scale - VAS), occurrence of nausea and vomiting (PONV), opioid consumption and side effects during 24 hours after surgery.

Conclusion:

The study aims to verify which anesthetic group provides less post-operative pain, less opioid consumption and greater patient well-being by not causing vomiting and nausea.

ELIGIBILITY:
Inclusion Criteria:Female patients aged between 18 and 80 years, ASA physical status I, II or III and undergoing unilateral surgery.

-

Exclusion Criteria: pregnant women, morbidly obese (BMI>40 kg/m²), patients with cognitive impairment or inability to communicate with the evaluator, coagulopathies, history of allergy to local anesthetics and patients with a history of chronic pain or drug addiction.

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | The visual analog scale (VAS) will be used to assess pain before surgery, in the PACU and after 24 hours, where 0 = no pain; 1-3 = mild pain; 4-6 = moderate pain; 7-10 = severe pain.
  To compare opioid consumption in patients undergoing breast surgery under general anesthesia associated with PECS II blockade or local anesthetic infiltration in the per- and post-operative periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nossa Senhora das Dores, Itabira, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cylwik J, Celinska-Spodar M, Buda N. Evaluation of the Efficacy of Pectoral Nerve-2 Block (PECS 2) in Breast Cancer Surgery. J Pers Med. 2023 Sep 24;13(10):1430. doi: 10.3390/jpm13101430. PMID 37888041
- [Background] Bakeer AH, Abdallah NM, Kamel MA, Abbas DN, Ragab AS. The impact of intravenous dexamethasone on the efficacy and duration of analgesia of paravertebral block in breast cancer surgery: a randomized controlled trial. J Pain Res. 2018 Dec 19;12:61-67. doi: 10.2147/JPR.S181788. eCollection 2019. PMID 30588080
- [Background] Bi Y, Ye Y, Zhu Y, Ma J, Zhang X, Liu B. The Effect of Ketamine on Acute and Chronic Wound Pain in Patients Undergoing Breast Surgery: A Meta-Analysis and Systematic Review. Pain Pract. 2021 Mar;21(3):316-332. doi: 10.1111/papr.12961. Epub 2020 Nov 13. PMID 33150677
- [Background] Badwe RA, Parmar V, Nair N, Joshi S, Hawaldar R, Pawar S, Kadayaprath G, Borthakur BB, Rao Thammineedi S, Pandya S, Balasubramanian S, Chitale PV, Neve R, Harris C, Srivastava A, Siddique S, Vanmali VJ, Dewade A, Gaikwad V, Gupta S. Effect of Peritumoral Infiltration of Local Anesthetic Before Surgery on Survival in Early Breast Cancer. J Clin Oncol. 2023 Jun 20;41(18):3318-3328. doi: 10.1200/JCO.22.01966. Epub 2023 Apr 6. PMID 37023374